CLINICAL TRIAL: NCT05050630
Title: A Perspective and Multicenter Phase II Trial of Tirelizumab Combined With R2-ICE Regimen (Rituximab, Lenalidomide, Ifosfamide, Carboplatin, Etoposide) in the Treatment of Refractory or Relapse DLBCL or HGBL
Brief Title: Phase II Trial of Tirelizumab Combined With R2-ICE Regimen in the Treatment of rrDLBCL/HGBL
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Affiliated Hospital to Academy of Military Medical Sciences (Other)
Collaborators: Peking University Cancer Hospital & Institute (Other); Cancer Institute and Hospital, Chinese Academy of Medical Sciences (Other)
Responsible Party: Principal Investigator, Huang Wenrong, Head of lymphoma and multiple myeloma department, Affiliated Hospital to Academy of Military Medical Sciences
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 307-947168-98
Record Dates: First submitted 2021-09-10; First posted 2021-09-20 (Actual); Last update posted 2021-09-20 (Actual); Status verified 2021-09

CONDITIONS: Age Range ≥16 Years, Gender Unlimited; Histopathology Confirmed Diffuse Large B-cell Lymphoma or High-grade B-cell Lymphoma; Received Prior First-line Chemotherapy for DLBCL or HGBL, Failed to Reach CR for Four Cycles, or Relapsed; At Least One Positive Lesion According to the 2014 Lugano Criteria for Hodgkin's and Non-Hodgkin's Lymphoma; ECOG Physical Status Score is 0-3; The Researchers Judged That Life Expectancy Was at Least Three Months; Understand and Voluntarily Sign Written Informed Consent
MeSH Terms: conditions — Lymphoma, Non-Hodgkin

STUDY DESIGN:
Intervention Model Description: All patients eligible for inclusion were treated with TR2-ICE：Rituximab 375 mg/m2 d0; Lenalidomide 25mg/d d1-10; Ifosfamide 5g/m2 d2; Carboplatin calculate according to AUC=5 (single dose ≤800 mg); Etoposide 100mg/m2 d1-3; Tirelizumab 200mg d6.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- TR2-ICE (Experimental): All patients eligible for inclusion were treated with TR2-ICE, and the first efficacy evaluation was conducted after the second course of treatment. If the patient can achieve complete response (CR), partial response (PR), and disease stability (SD), the clinical benefit is considered, and the TR2-ICE treatment regimen is continued. The second efficacy assessment was performed after the 4th course of treatment. If patients achieved complete response (CR) or partial response (PR) compared to baseline, the clinical treatment was considered effective and the TR2-ICE treatment regimen was continued. After the completion of six courses of induction chemotherapy, an end-of-course assessment was performed. Patients with CR and PR can choose to undergo autologous hematopoietic stem cell transplantation consolidation therapy, or lenalidomide or Tirelarizin monotherapy or both combination maintenance therapy.
  Interventions: Drug: TR2-ICE

INTERVENTIONS:
Drug: TR2-ICE — Rituximab 375 mg/m2 d0; Lenalidomide 25mg/d d1-10; Ifosfamide 5g/m2 d2; Carboplatin calculate according to AUC=5 (single dose ≤800 mg); Etoposide 100mg/m2 d1-3; Tirelizumab 200mg d6.

SUMMARY:
This study was a prospective, multi-center, single-arm, Phase II clinical study. Compared with the literature data, objective response rate (ORR) and complete response rate (CR) were the primary endpoint, and 1-year and 2-year progression-free survival (PFS) and 2-year overall survival (OS) were the secondary endpoint. To evaluate the efficacy and safety of TR2-ICE sequential Tirelarizin, lenalidomide alone, or both maintenance therapy in the rescue of patients with relapsed and refractory diffuse large B or high-grade B-cell lymphoma.

DETAILED DESCRIPTION:
All patients eligible for inclusion were treated with TR2-ICE, and the first efficacy evaluation was conducted after the second course of treatment. If the patient can achieve complete response (CR), partial response (PR), and disease stability (SD), the clinical benefit is considered, and the TR2-ICE treatment regimen is continued. The second efficacy assessment was performed after the 4th course of treatment. If patients achieved complete response (CR) or partial response (PR) compared to baseline, the clinical treatment was considered effective and the TR2-ICE treatment regimen was continued. After the completion of six courses of induction chemotherapy, an end-of-course assessment was performed. Patients with CR and PR can choose to undergo autologous hematopoietic stem cell transplantation consolidation therapy, or lenalidomide or Tirelarizin monotherapy or both combination maintenance therapy. If patients still had SD after four courses of treatment or PD at any time during the study, they were dropped out of the study and given salvage therapy.

ELIGIBILITY:
Inclusion Criteria:

1. Age range ≥16 years old, no gender limitation;
2. Diffuse large B-cell lymphoma or high-grade B-cell lymphoma (HGBL) was confirmed by histopathology.
3. Have received prior first-line chemotherapy for DLBCL or HGBL, failed to reach CR in four cycles, or relapsed.
4. At least one positive lesion under 18F-deoxyglucose (18FDG) positron emission computed tomography (PET-CT) according to the 2014 Lugano criteria for Hodgkin's and non-Hodgkin's lymphoma;
5. ECOG physical status score is 0-3;
6. At the time of screening, laboratory tests met the following criteria, unless the investigator could determine that lymphoma was the cause (no corrective and supportive treatment for the parameters described below was performed within 2 weeks prior to evaluation) : (1) Routine blood test: Hemoglobin (Hb) ≥90g/L, absolute neutrophil (ANC) ≥1.5×109/L, platelet count (PLT) ≥90×109/L; (2) biochemical examination: serum creatinine (Cr) ≤1.5× upper limit of normal value (ULN), creatinine clearance rate > 50ml/min (Cockcroft formula); Total bilirubin (TBIL) ≤1.5×ULN; Alanine aminotransferase (ALT) and aspartate aminotransferase (AST) ≤2.5×ULN (liver metastasis: ≤5ULN).
7. Life expectancy was at least three months, the researchers judged;
8. Understand and voluntarily sign written informed consent.

Exclusion Criteria:

1. With central nervous system metastasis or piameningeal metastasis;
2. Prior organ transplant;
3. Previous or current combination of other malignant tumors, except adequately treated basal cell carcinoma or squamous cell carcinoma of the skin, carcinoma in situ of the cervix;
4. Patients who have been treated with PD-1 inhibtor before;
5. History of severe allergy to antibody drugs;
6. Those with active immune diseases, such as systemic lupus erythematosus;
7. Uncontrolled or significant cardiovascular disease, including: (1) New York Heart Association (NYHA) class II or higher congestive heart failure, unstable angina, myocardial infarction, or arrhythmia requiring treatment, or left ventricular ejection fraction (LVEF) <50% at the time of screening within 6 months prior to initial administration of the study drug; (2) primary cardiomyopathy (such as dilated cardiomyopathy, hypertrophic cardiomyopathy, arrhythmogenic right ventricular cardiomyopathy, restricted cardiomyopathy, unshaped cardiomyopathy); (3) clinically significant prolonged history of QTc interval, or screening QTc interval >470ms for women and >450ms for men; (4) symptomatic coronary heart disease requiring drug treatment during screening period; (5) Other cardiovascular diseases deemed unsuitable for inclusion by the investigator.
8. A history of severe interstitial lung disease (ILD), such as pulmonary fibrosis, or baseline chest CT or MRI showing evidence of ILD;
9. Clinically significant gastrointestinal abnormalities that may affect drug intake, transport or absorption (such as inability to swallow, chronic diarrhea, intestinal obstruction, etc.), or total gastrectomy;
10. High-risk surgery for vital organs or poor healing of other surgical wounds as determined by the investigator 6 weeks prior to screening;
11. Active infection or active or uncontrolled HBV, HCV infection, HIV/AIDS (Acquired Immune Deficiency Syndrome) or other serious infectious diseases (including: active infection requiring systemic treatment; HBV/HCV/HIV qualitative detection is preferred, quantitative detection is required; HBV DNA can be included after treatment to turn negative);
12. Any mental or cognitive impairment that may limit their understanding of informed consent, performance of informed consent, and compliance with the study;
13. Drug and alcohol abuse;
14. Women of reproductive age who are unwilling or unable to use an effective method of contraception during the entire treatment period of the trial and within 12 weeks of the last Tirelizu administration or within 12 months of the last rituximab administration, whichever is the latest [women of reproductive age include: Any woman who has menstruated and has not undergone successful artificial sterilization (hysterectomy, bilateral tubal ligation or bilateral oophorectomy) or has not been menopausal], is pregnant or breastfeeding;
15. Other conditions that the investigator considers inappropriate for participation in the study.

Min Age: 16 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 73 (Estimated)
Dates: Start 2021-08-01 (Actual); Primary Completion 2022-07-30 (Estimated); Study Completion 2023-07-30 (Estimated)

PRIMARY OUTCOMES:
Main purpose | Enrollment is expected to last for one year, followed up for two years.
  Compared with the literature data, objective response rate (ORR) and complete response rate (CR) were the primary endpoint

CONTACTS AND LOCATIONS:
Locations (1):
- Hospital 307, Beijing, Beijing Municipality, China

IPD SHARING:
Plan to Share IPD: No